CLINICAL TRIAL: NCT01756898
Title: A Multicenter, Randomized, Placebo-Controlled, Double-Blind, Parallel-group Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of ASB17061 Capsules in Adult Subjects With Atopic Dermatitis
Brief Title: Study to Evaluate the Efficacy, Safety and Pharmacokinetics of ASB17061 Capsules in Adult Subjects With Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ASBI 704
Record Dates: First submitted 2012-11-09; First posted 2012-12-28 (Estimated); Results first posted 2021-02-16 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-01

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Low dose ASB17061 (Experimental): Oral administration of low dose ASB17061 taken once daily for 28 consecutive days.
  Interventions: Drug: 5 mg ASB17061
- Middle dose ASB17061 (Experimental): Oral administration of middle dose ASB17061 taken once daily for 28 consecutive days.
  Interventions: Drug: 10 mg ASB17061
- High dose ASB17061 (Experimental): Oral administration of high dose ASB17061 taken once daily for 28 consecutive days.
  Interventions: Drug: 20 mg ASB17061
- Placebo (Placebo Comparator): Oral administration of placebo taken once daily for 28 consecutive days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 5 mg ASB17061 — Oral administration of 5 mg ASB17061 taken once daily for 28 consecutive days.
  Arms: Low dose ASB17061
Drug: Placebo — Oral administration of placebo taken once daily for 28 consecutive days.
  Arms: Placebo
Drug: 10 mg ASB17061 — Oral administration of 10 mg ASB17061 taken once daily for 28 consecutive days.
  Arms: Middle dose ASB17061
Drug: 20 mg ASB17061 — Oral administration of 20 mg ASB17061 taken once daily for 28 consecutive days.
  Arms: High dose ASB17061

SUMMARY:
The purpose of this research study is to gather scientific information about the effectiveness of the study drug, ASB17061 capsules, when compared to placebo in adult subjects with atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects ages 18 to 65 years
* A diagnosis of atopic dermatitis (AD)
* An Investigator's Global Assessment (IGA) score of 2 or higher and AD affecting at least 5% of total Body Surface Area (BSA)
* Other than active AD, in good health with no medical condition that may jeopardize the safety of the subject or impact the validity of the study results
* Subjects must be practicing acceptable birth control methods

Exclusion Criteria:

* Taking systemic immunosuppressive therapy within 3 months prior to screening or systemic (cortico) steroid therapy within 4 weeks prior to screening
* Use of phototherapy or tanning beds within 6 weeks of screening
* Presence of a clinically significant disorder involving gastrointestinal, renal, hepatic, neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic, psychiatric, or cardiovascular disease or any other condition, which will jeopardize the safety of the subject or impact the validity of the study results
* Female subjects who are pregnant or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Actual)
Dates: Start 2012-11-28 (Actual); Primary Completion 2014-01-14 (Actual); Study Completion 2014-01-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (38):
- United States (38):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Rogers, Arkansas
  - Encino, California
  - Fremont, California
  - San Diego, California
  - Temecula, California
  - Denver, Colorado
  - Miami, Florida
  - Miramar, Florida
  - Saint Augustine, Florida
  - South Tampa, Florida
  - Tampa, Florida
  - Savannah, Georgia
  - Boise, Idaho
  - Overland Park, Kansas
  - Crowley, Louisiana
  - Bay City, Michigan
  - Clinton Township, Michigan
  - Fort Gratiot, Michigan
  - Berlin, New Jersey
  - Verona, New Jersey
  - Stony Brook, New York
  - Raleigh, North Carolina
  - Sylvania, Ohio
  - Lake Oswego, Oregon
  - Portland, Oregon
  - Johnston, Rhode Island
  - Arlington, Texas
  - College Station, Texas
  - Pflugerville, Texas
  - San Antonio, Texas
  - Webster, Texas
  - Draper, Utah
  - West Jordan, Utah
  - Henrico, Virginia
  - Norfolk, Virginia
  - Spokane, Washington

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 370 participants who met all inclusion criteria and no exclusion criteria were enrolled in the study at 42 clinic sites in the United States of America.
Pre-assignment Details: Adult male and female subjects with active atopic dermatitis (AD) were enrolled in this study.
Groups:
- Placebo: Participants with atopic dermatitis were randomized to receive a placebo.
- ASB17061 5 mg Low Dose: Participants with atopic dermatitis were randomized to receive ASB17061 low dose (5 mg).
- ASB17061 10 mg Middle Dose: Participants with atopic dermatitis were randomized to receive ASB17061 medium dose (10 mg).
- ASB17061 20 mg High Dose: Participants with atopic dermatitis were randomized to receive ASB17061 high dose (20 mg).
Period: Overall Study
Arm/Group | Placebo | ASB17061 5 mg Low Dose | ASB17061 10 mg Middle Dose | ASB17061 20 mg High Dose
Started | 92 | 92 | 93 | 93
Completed | 73 | 73 | 76 | 77
Not Completed | 19 | 19 | 17 | 16
Not completed — Adverse Event | 7 | 1 | 0 | 0
Not completed — Lack of Efficacy | 4 | 7 | 6 | 6
Not completed — Lost to Follow-up | 2 | 4 | 2 | 3
Not completed — Protocol Violation | 1 | 2 | 2 | 1
Not completed — Withdrew Consent | 5 | 3 | 5 | 6
Not completed — Other | 0 | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were assessed in the Intent-to-Treat (ITT) population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | ASB17061 5 mg Low Dose | ASB17061 10 mg Middle Dose | ASB17061 20 mg High Dose | Total
Number analyzed (Participants) | 91 | 90 | 92 | 93 | 366
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.0 (13.34) | 36.9 (14.34) | 37.1 (14.82) | 39 (13.71) | 37.7 (14.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 68 | 60 | 72 | 260
  Male | 31 | 22 | 32 | 21 | 106
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 19 | 21 | 22 | 84
  Not Hispanic or Latino | 69 | 71 | 71 | 71 | 282
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 6 | 2 | 6 | 6 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 26 | 25 | 21 | 23 | 95
  White | 55 | 58 | 62 | 60 | 235
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 5 | 3 | 4 | 16
Region of Enrollment [Number; unit: participants]
  United States | 91 | 90 | 92 | 93 | 366

OUTCOME MEASURES:

1. Primary Outcome: Number of Investigator's Global Assessment (IGA) Responders at Day 29 Following Treatment With ASB17061 Capsules or Placebo in Adults With Atopic Dermatitis
Description: Participants with an IGA score of 0 or 1 were considered IGA responders. The investigator provided an overall assessment of disease severity using the IGA, which consists of a 6-point scale from a minimum of 0 and a maximum of 6. Higher scores indicate a worse outcome and lower scores indicate a better outcome. (0 = clear; 1 = almost clear; 2 = mild disease; 3 = moderate disease, 4 = severe disease; and 5 = very severe disease).
Time Frame: Baseline up to 29 days after initial dose.
Population: The Intent-to-Treat population, last observation carried forward (LOCF) was used to assess IGA.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | ASB17061 5 mg Low Dose | ASB17061 10 mg Middle Dose | ASB17061 20 mg High Dose
Number analyzed (Participants) | 91 | 90 | 92 | 93
Participants | 20 | 21 | 19 | 18

2. Primary Outcome: Number of Investigator's Global Assessment (IGA) Responders By Subgroup at Day 29 Following Treatment With ASB17061 Capsules or Placebo in Adults With Atopic Dermatitis
Description: Participants with an IGA score of 0 or 1 were considered IGA responders. The investigator provided an overall assessment of disease severity using the IGA which consists of a 6-point scale from the minimum of 0 to a maximum of 6. Higher scores indicate increasing severity.. (0 = clear; 1 = almost clear; 2 = mild disease; 3 = moderate disease, 4 = severe disease; and 5 = very severe disease) and an overall assessment of the disease severity of the entire body using the Eczema Area and Severity Index (EASI). A composite index, the EASI has a minimum score of 0 (clear) and a maximum score of 72 (very severe); A value less than 15 indicates less severe, and 15 or greater indicates more severe. Lichenification was evaluated on a scale of 0 (none) as the minimum to 3 (severe) as the maximum, and the score of each body region was summed (0 to 12). A percent body surface area (BSA) involved less than 15 is less severe and 15 or greater more severe.
Time Frame: Baseline up to 29 days after initial dose.
Population: The Intent-to-Treat population, last observation carried forward (LOCF) was used to assess IGA by subgroup.
Measure: Number; unit: participants
Arm/Group | Placebo | ASB17061 5 mg Low Dose | ASB17061 10 mg Middle Dose | ASB17061 20 mg High Dose
Number analyzed (Participants) | 91 | 90 | 92 | 93
participants
  Male: number analyzed (Participants) | 31 | 22 | 32 | 21
  Male | 1 | 3 | 7 | 7
  Female: number analyzed (Participants) | 60 | 68 | 60 | 72
  Female | 19 | 18 | 12 | 11
  White: number analyzed (Participants) | 55 | 58 | 62 | 60
  White | 13 | 12 | 14 | 13
  Black or African American: number analyzed (Participants) | 26 | 25 | 21 | 23
  Black or African American | 6 | 6 | 4 | 4
  Other: number analyzed (Participants) | 10 | 7 | 9 | 10
  Other | 1 | 3 | 1 | 1
  Baseline EASI score <15: number analyzed (Participants) | 63 | 66 | 70 | 70
  Baseline EASI score <15 | 18 | 20 | 18 | 17
  Baseline EASI score ≥15: number analyzed (Participants) | 28 | 24 | 22 | 23
  Baseline EASI score ≥15 | 2 | 1 | 1 | 1
  Baseline Lichenification severity 0-3: number analyzed (Participants) | 35 | 30 | 37 | 31
  Baseline Lichenification severity 0-3 | 15 | 9 | 10 | 8
  Baseline Lichenification severity 4-12: number analyzed (Participants) | 56 | 60 | 55 | 62
  Baseline Lichenification severity 4-12 | 5 | 12 | 9 | 10
  Baseline % BSA involved <15%: number analyzed (Participants) | 48 | 59 | 59 | 55
  Baseline % BSA involved <15% | 16 | 19 | 16 | 15
  Baseline % BSA involved ≥15%: number analyzed (Participants) | 43 | 31 | 33 | 38
  Baseline % BSA involved ≥15% | 4 | 2 | 3 | 3
  Baseline IGA score = 2: number analyzed (Participants) | 22 | 18 | 20 | 23
  Baseline IGA score = 2 | 9 | 9 | 10 | 8
  Baseline IGA score = 3: number analyzed (Participants) | 47 | 50 | 52 | 47
  Baseline IGA score = 3 | 11 | 12 | 8 | 9
  Baseline IGA score = 4 or 5: number analyzed (Participants) | 22 | 22 | 20 | 23
  Baseline IGA score = 4 or 5 | 0 | 0 | 1 | 1
  Baseline IGA score = 3, 4, or 5: number analyzed (Participants) | 69 | 72 | 72 | 70
  Baseline IGA score = 3, 4, or 5 | 11 | 12 | 9 | 10
  Allergic rhinitis/Asthma absent: number analyzed (Participants) | 44 | 48 | 57 | 49
  Allergic rhinitis/Asthma absent | 10 | 10 | 8 | 13
  Allergic rhinitis/Asthma present: number analyzed (Participants) | 47 | 42 | 35 | 44
  Allergic rhinitis/Asthma present | 10 | 11 | 11 | 5
  Baseline Immunoglobulin (IgE) <100 IU/mL: number analyzed (Participants) | 37 | 35 | 44 | 38
  Baseline Immunoglobulin (IgE) <100 IU/mL | 14 | 10 | 13 | 11
  Baseline Immunoglobulin (IgE) ≥100 IU/mL: number analyzed (Participants) | 53 | 54 | 47 | 54
  Baseline Immunoglobulin (IgE) ≥100 IU/mL | 6 | 10 | 6 | 7

3. Secondary Outcome: Mean Change From Baseline in Eczema Area and Severity Index Score (EASI) Following Treatment With ASB17061 Capsules or Placebo in Adult Participants With Atopic Dermatitis at Day 29
Description: The investigator provided an overall assessment of the disease severity of the entire body using the EASI. A composite index, the EASI has a minimum score of 0 (clear) and a maximum score of 72 (very severe); with a negative value indicating decreasing severity of eczema compared to baseline and a decreasing change in the EASI score. A negative value is an indication of a decrease in individual scores.
Time Frame: Baseline up to 29 days after initial dose.
Population: The Intent-to-Treat population, last observation carried forward (LOCF) was used to assess EASI.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | ASB17061 5 mg Low Dose | ASB17061 10 mg Middle Dose | ASB17061 20 mg High Dose
Number analyzed (Participants) | 91 | 90 | 92 | 93
Units on a scale
  Baseline | 12.6 (11.2) | 12.2 (9.67) | 11.2 (9.12) | 11.7 (9.96)
  Day 29 | -3.43 (7.96) | -3.24 (7.45) | -3.51 (6.75) | -2.75 (4.77)

4. Secondary Outcome: Mean Change From Baseline in The Percentage of Body Surface Area (BSA) Involved Following Treatment With ASB17061 Capsules or Placebo in Adult Participants With Atopic Dermatitis at Day 29
Description: Participants' body surface area affected by atopic dermatitis was assessed for the change in percentage after treatment. A negative value indicates a decrease in the percent of body surface area (BSA) involved. A negative value is an indication of a decrease in individual scores.
Time Frame: Baseline up to 29 days after initial dose.
Population: The Intent-to-Treat population, last observation carried forward (LOCF) was used to assess the percent Body Surface Area.
Measure: Mean (Standard Deviation); unit: Percentage of BSA
Arm/Group | Placebo | ASB17061 5 mg Low Dose | ASB17061 10 mg Middle Dose | ASB17061 20 mg High Dose
Number analyzed (Participants) | 91 | 90 | 92 | 93
Percentage of BSA
  Baseline | 21.0 (20.87) | 19.6 (21.96) | 18.5 (19.00) | 18.1 (17.29)
  Day 29 | -3.59 (7.69) | -2.99 (9.44) | -2.95 (6.23) | -3.27 (6.50)

5. Secondary Outcome: Mean Change From Baseline in Pruritus Score Following Treatment With ASB17061 Capsules or Placebo in Adult Participants With Atopic Dermatitis at Day 29
Description: Participants assessed the overall intensity of pruritus using a 4-point scale with 0 as the minimum and 3 as the maximum. (0 = absent; 1 = mild; 2 = moderate; and 3 = severe) A negative value indicates a decreasing change in the pruritus score. A negative value is an indication of a decrease in individual scores.
Time Frame: Baseline up to 29 days after initial dose.
Population: The Intent-to-Treat population, last observation carried forward (LOCF) was used to assess pruritus score.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | ASB17061 5 mg Low Dose | ASB17061 10 mg Middle Dose | ASB17061 20 mg High Dose
Number analyzed (Participants) | 91 | 90 | 92 | 93
Units on a scale
  Baseline | 2.3 (0.74) | 2.4 (0.68) | 2.2 (0.72) | 2.5 (0.64)
  Day 29 | -0.75 (1.00) | -0.80 (0.97) | -0.72 (1.03) | -0.76 (0.90)

6. Secondary Outcome: Mean Change From Baseline in Insomnia Score Following Treatment With ASB17061 Capsules or Placebo in Adult Participants With Atopic Dermatitis at Day 29
Description: Participants assessed the extent of their insomnia using an 11-point scale ranging from the minimum, 0 (no insomnia) to the maximum, 10 (severe insomnia). A negative value indicates a decreasing change in the insomnia score. A negative value is an indication of a decrease in individual scores.
Time Frame: Baseline up to 29 days after initial dose.
Population: The Intent-to-Treat population, last observation carried forward (LOCF) was used to assess the insomnia score.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | ASB17061 5 mg Low Dose | ASB17061 10 mg Middle Dose | ASB17061 20 mg High Dose
Number analyzed (Participants) | 91 | 90 | 92 | 93
Units on a scale
  Baseline | 4.0 (3.13) | 3.9 (3.09) | 3.7 (3.30) | 3.6 (2.76)
  Day 29 | -1.10 (2.69) | -1.06 (2.76) | -1.20 (3.02) | -0.97 (2.20)

7. Secondary Outcome: Plasma Concentrations of ASB17061 and ASB17584 Over Time Following Treatment With ASB17061 Capsules in Adult Participants With Atopic Dermatitis
Time Frame: Baseline (Day 1 Predose) up to Day 8, Day 15, and Day 22 at 0 to 2.5 hours, 2.5 to 5 hours, 5 to 10 hours, up to Day 29 at 24-32 hours postdose.
Population: The Pharmacokinetic (PK) sample analyses were performed on the PK Population. Only plasma samples from active participants were analyzed for ASB17061 and ASB17584 concentrations.
Measure: Mean (Standard Deviation); unit: ng/ML
Arm/Group | ASB17061 5 mg Low Dose | ASB17061 10 mg Middle Dose | ASB17061 20 mg High Dose
Number analyzed (Participants) | 92 | 93 | 93
ng/ML
  Predose ASB17061: number analyzed (Participants) | 91 | 91 | 93
  Predose ASB17061 | NA (NA) — Not Detected (less than 0.5 ng/mL) | NA (NA) — Not Detected (less than 0.5 ng/mL) | NA (NA) — Not Detected (less than 0.5 ng/mL)
  0 to 2.5 hours ASB17061: number analyzed (Participants) | 75 | 80 | 92
  0 to 2.5 hours ASB17061 | 24.4 (18.7) | 48.3 (51.4) | 89.6 (78.6)
  2.5 to 5 hours ASB17061: number analyzed (Participants) | 85 | 89 | 90
  2.5 to 5 hours ASB17061 | 18.3 (13.7) | 33.3 (24.9) | 72.7 (48.2)
  5 to 10 hours ASB17061: number analyzed (Participants) | 70 | 75 | 83
  5 to 10 hours ASB17061 | 8.03 (9.15) | 18.0 (20.6) | 38.8 (55.2)
  Day 29 (24-32 hours) ASB17061: number analyzed (Participants) | 26 | 42 | 55
  Day 29 (24-32 hours) ASB17061 | 3.07 (6.30) | 5.32 (15.2) | 3.35 (8.27)
  Predose ASB17584: number analyzed (Participants) | 91 | 91 | 93
  Predose ASB17584 | NA (NA) — Not Detected (less than 0.5 ng/mL) | NA (NA) — Not Detected (less than 0.5 ng/mL) | NA (NA) — Not Detected (less than 0.5 ng/mL)
  0 to 2.5 hours ASB17584: number analyzed (Participants) | 67 | 66 | 88
  0 to 2.5 hours ASB17584 | 9.21 (7.63) | 18.1 (17.1) | 27.3 (25.2)
  2.5 to 5 hours ASB17584: number analyzed (Participants) | 81 | 88 | 89
  2.5 to 5 hours ASB17584 | 7.50 (5.60) | 14.4 (13.0) | 30.7 (21.3)
  5 to 10 hours ASB17584: number analyzed (Participants) | 67 | 73 | 83
  5 to 10 hours ASB17584 | 2.98 (3.67) | 6.29 (6.16) | 15.1 (20.5)
  Day 29 (24-32 hours) ASB17584: number analyzed (Participants) | 12 | 21 | 37
  Day 29 (24-32 hours) ASB17584 | 2.40 (4.21) | 2.31 (3.11) | 2.11 (4.24)

8. Secondary Outcome: Minimum Observed Plasma Concentration (Cmin) of ASB17061 and ASB17584 Following Treatment With ASB17061 Capsules in Adult Participants With Atopic Dermatitis
Description: The minimum observed plasma drug concentration (Cmin) of ASB17061 and ASB17584 in the 4-week Treatment Period were estimated from the actual dosing records.
Time Frame: as for outcome 7
Population: The Cmin was assessed in the Efficacy Evaluable (EE) Population.
Measure: Mean (Standard Deviation); unit: ng/ML
Arm/Group | ASB17061 5 mg Low Dose | ASB17061 10 mg Middle Dose | ASB17061 20 mg High Dose
Number analyzed (Participants) | 71 | 72 | 82
ng/ML
  Cmin ASB17061 | 0.88 (2.09) | 1.34 (0.94) | 2.43 (2.44)
  Cmin ASB17584 | 0.58 (0.76) | 0.97 (0.69) | 1.82 (1.58)

9. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of ASB17061 and ASB17584 Following Treatment With ASB17061 Capsules in Adult Subjects With Atopic Dermatitis
Description: Pharmacokinetic (PK) metrics of ASB17061 and ASB17584 maximum observed plasma drug concentration (Cmax) in the 4-week Treatment Period were estimated from the individual PK parameters and the actual dosing records.
Time Frame: as for outcome 7
Population: The Cmax was assessed in the Efficacy Evaluable (EE)Population.
Measure: Mean (Standard Deviation); unit: ng/ML
Arm/Group | ASB17061 5 mg Low Dose | ASB17061 10 mg Middle Dose | ASB17061 20 mg High Dose
Number analyzed (Participants) | 71 | 72 | 82
ng/ML
  Cmax ASB17061 | 33.82 (13.67) | 67.60 (19.39) | 134.90 (53.94)
  Cmax ASB17584 | 11.27 (4.24) | 22.25 (8.79) | 42.73 (15.36)

10. Secondary Outcome: Average Plasma Concentration (Cavg) of ASB17061 and ASB17584 Following Treatment With ASB17061 Capsules in Adult Participants With Atopic Dermatitis
Description: The average plasma drug concentration (Cmin) of ASB17061 and ASB17584 in the 4-week Treatment Period were estimated from the actual dosing records.
Time Frame: Baseline up to Predose, up to 0 to 2.5 hours, up to 2.5 to 5 hours, up to 5 to 10 hours, up to Day 29 (24-32 hours).
Population: The Cavg was analyzed in the Efficacy Evaluable Population.
Measure: Mean (Standard Deviation); unit: ng/ML
Arm/Group | ASB17061 5 mg Low Dose | ASB17061 10 mg Middle Dose | ASB17061 20 mg High Dose
Number analyzed (Participants) | 71 | 72 | 82
ng/ML
  Cavg ASB17061 | 5.59 (3.57) | 11.04 (4.21) | 21.88 (10.30)
  Cavg ASB17584 | 2.16 (1.21) | 4.18 (2.04) | 8.30 (3.84)

11. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAE) Following Treatment With ASB17061 Capsules or Placebo in Adult Participants With Atopic Dermatitis
Description: A treatment-emergent adverse event (TEAE) was defined as an AE that emerges during treatment, having been absent at pre-treatment; or reemerges during treatment, having been present at baseline but stopped prior to treatment; or worsens in severity during treatment after initiating the study drug.
Time Frame: Baseline up to Day 57 follow-up visit post dose.
Population: Treatment-emergent adverse events (TEAEs) were assessed in the Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | ASB17061 5 mg Low Dose | ASB17061 10 mg Middle Dose | ASB17061 20 mg High Dose
Number analyzed (Participants) | 92 | 92 | 93 | 93
Participants
  Bronchitis | 0 | 2 | 3 | 1
  Influenza | 1 | 0 | 4 | 0
  Nasopharyngitis | 4 | 7 | 7 | 6
  Sinusitis | 1 | 2 | 0 | 1
  Upper respiratory tract infection | 4 | 3 | 4 | 2
  Urinary tract infection | 0 | 3 | 2 | 2
  Abdominal pain | 2 | 0 | 1 | 2
  Abdominal pain upper | 1 | 1 | 2 | 2
  Constipation | 0 | 2 | 0 | 1
  Diarrhea | 4 | 2 | 4 | 5
  Dyspepsia | 0 | 2 | 0 | 0
  Flatulence | 2 | 3 | 2 | 0
  Nausea | 2 | 1 | 2 | 4
  Vomiting | 2 | 2 | 5 | 2
  Dermatitis atopic | 3 | 8 | 5 | 3
  Dermatitis contact | 2 | 0 | 0 | 0
  Eczema | 0 | 1 | 2 | 1
  Pruritis | 1 | 0 | 2 | 2
  Urticaria | 0 | 0 | 3 | 0
  Headache | 4 | 9 | 6 | 9
  Somnolence | 1 | 0 | 3 | 0
  Aspartate aminotransferase increased | 2 | 0 | 1 | 0
  Blood creatine phosphokinase increased | 6 | 0 | 4 | 2
  Blood testosterone decreased | 3 | 0 | 0 | 1
  Hepatic enzyme increased | 2 | 0 | 0 | 0
  White blood cell count increased | 0 | 0 | 0 | 2
  Cough | 1 | 2 | 1 | 2
  Oropharyngeal pain | 1 | 2 | 3 | 0
  Rhinorrhea | 2 | 1 | 0 | 0
  Myalgia | 1 | 3 | 1 | 2
  Fatigue | 2 | 2 | 1 | 0
  Arthropod bite | 0 | 0 | 2 | 0
  Ligament sprain | 0 | 0 | 2 | 0
  Insomnia | 0 | 2 | 2 | 0
  Polyuria | 0 | 2 | 0 | 0
  Ovarian cyst | 0 | 2 | 0 | 0
  Hypertension | 0 | 0 | 2 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 12 weeks after the initial dose.
Description: A treatment-emergent adverse event (TEAE) was defined as an AE that emerges during treatment, having been absent at pre-treatment; or reemerges during treatment, having been present at baseline but stopped prior to treatment; or worsens in severity during treatment after initiating the study drug.
Arm/Group | Placebo | ASB17061 5 mg Low Dose | ASB17061 10 mg Middle Dose | ASB17061 20 mg High Dose
All-Cause Mortality (participants affected / at risk) | 0/92 | 0/92 | 0/93 | 0/93
Serious Adverse Events (participants affected / at risk) | 0/92 | 1/92 | 0/93 | 0/93
Other Adverse Events (participants affected / at risk) | 44/92 | 51/92 | 54/93 | 45/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=92) | ASB17061 5 mg Low Dose (N=92) | ASB17061 10 mg Middle Dose (N=93) | ASB17061 20 mg High Dose (N=93)
Bilateral Clubfoot (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=92) | ASB17061 5 mg Low Dose (N=92) | ASB17061 10 mg Middle Dose (N=93) | ASB17061 20 mg High Dose (N=93)
Nasopharyngitis (Infections and infestations) | 13 | 25 | 24 | 17
Diarrhea (Gastrointestinal disorders) | 10 | 15 | 16 | 10
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 8 | 11 | 10 | 7
Headache (Nervous system disorders) | 6 | 9 | 10 | 9
Blood creatine phosphokinase increased (Investigations) | 13 | 1 | 7 | 8
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 4 | 8 | 5 | 5
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 5 | 4 | 2 | 7
General disorders and administration site conditions (General disorders) | 5 | 3 | 3 | 2
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 1 | 1 | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No